CLINICAL TRIAL: NCT00631683
Title: Use of Flo-Trac/Vigileo (TM) for Hemodynamic Monitoring During Discontinuation From Mechanical Ventilation
Brief Title: Assessment of Hemodynamic Changes During Weaning From Mechanical Ventilation With Flo-Trac Vigileo (TM) Monitor.
Status: Withdrawn | Type: Observational
Why Stopped: Terms for legal agreements between institution and Sponsor could not be made.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC-MS-07-0368
Record Dates: First submitted 2008-02-22; First posted 2008-03-10 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MICU-1: Mechanically ventilated patients who are about to start a weaning trial at the medical intensive care unit of Memorial Hermann Hospital.

SUMMARY:
Failure to wean from mechanical ventilation (failure to get the patients off the breathing machine) is associated with prolonged stay in the intensive care unit and increased risk of death. Some patients have difficulty successfully getting off the ventilator and breathing on their own. Usually this difficulty is due to lung problems. But sometimes it is due to heart problems, or heart failure. To improve a patient's chances of successfully getting off the ventilator early, it is helpful to the doctors to know if patient has heart failure and to measure how severe. With the new monitoring system being studied here, doctors may be able to detect and measure heart failure more easily.

A new monitor (Vigileo TM) that is connected with a specific cable (Flo-TracTM) to a catheter that is inside the patient's artery (arterial line) has lately been developed. This monitor can estimate the amount of blood that the heart is pumping per minute, known as cardiac output. The heart is supposed to pump blood harder when a patient is being weaned from the breathing machine. With the above mentioned monitor, we hope to detect those patients whose hearts are weak and are not pumping as hard as they should.

DETAILED DESCRIPTION:
In the process of liberation or discontinuation from mechanical ventilation (also commonly referred as "weaning") the goal is to achieve spontaneous breathing and ultimately extubation. Weaning failure occurs in up to 25% of patients who meet criteria for weaning, especially in those with underlying COPD or heart failure (1). Weaning failure is well known to prolong intensive care unit (ICU) stay, and to increase morbidity and mortality in critically ill patients. Early identification and treatment of causes of weaning failure is of paramount importance to improve outcome in difficult to wean patients.

Although respiratory system failure is the most common cause of weaning failure, occult cardiovascular insufficiency occurs very often in critically ill patients, and it can contribute to, or be the only cause of weaning failure in many patients (2). Recognition of cardiovascular origin of weaning failure is crucial since the use of vasodilators and/or diuretics may result in successful weaning (1).

Cardiovascular instability during liberation from mechanical ventilation was first described more than 30 years ago by Beach et al (3) in post-operative cardiac surgery patients. Since then, a few other studies have described the hemodynamic changes both in patients who underwent successful and unsuccessful weaning form mechanical ventilation (1,4,5,6,7). Lemaire et al. (4) emphasized the use of a pulmonary artery catheter as the "gold standard" to detect left ventricular dysfunction during spontaneous breathing trial (SBT). They reported a markedly increased in pulmonary artery occlusion pressure (PAOP) in patients who were suffering from COPD or heart failure who failed to wean from mechanical wentilation. Jubran et al. (5) reported an increase in PAOP, decreased mixed venous oxygen saturation (SvO2) and an increase in the oxygen extraction ratio in a group of patients who failed to wean from mechanical ventilation. In contrast, De Backer et al. (6) described an increase in cardiac index in a group of patients who were successfully weaned after cardiac surgery. A recently published study by Frazier et al. (7) corroborated previous data by comparing the hemodynamic changes between a group of patients who were successfully weaned and a group of patients who failed to wean from mechanical ventilation. The cardiac output and stroke volume were estimated by the differential Fick partial rebreathing technique, with carbon dioxide as the indicator substance. The group of patients who were successfully weaned had a statistical significant increase in both stroke volume and cardiac index, unlike the group that failed weaning.

The physiologic changes that explain the above mentioned findings in hemodynamic parameters during weaning are complex and not fully understood (1). It is well known that weaning can place an excessive burden on the heart and it can be considered a form of "exercise" (2). As studied by exercise physiologists, the increase in oxygen consumption during exercise in healthy individuals is matched both by an increase in cardiac output and oxygen extraction. In patients with overt heart failure, the increase in cardiac output is inadequate, and the predominant response constitutes and increase in oxygen extraction. Return to spontaneous breathing induces alteration in intrathoracic pressures that influence cardiovascular function, producing, among other changes, an increase in venous return. Other postulated physiologic changes include increase sympathetic tone, weaning-induced myocardial ischemia and increased ventricular interdependence (2).

The recognition of cardiac origin of weaning failure is of vital importance. Unfortunately, the clinical signs of patients who fail weaning because of acute heart failure (tachypnea, tachycardia, anxiety, etc) are often difficult to distinguish from signs of respiratory failure. Reliable bedside minimally invasive monitoring tools and tests need to be developed to help the clinician in identifying these patients and help titrate cardiovascular therapies during weaning trials. Currently, the list of such tools is short and the validity of each technique in different situations is unknown (2).

Cardiovascular dysfunction may be the missing piece in predicting weaning success. Cardiovascular monitoring can be useful in identifying and managing patients who fail to wean due to lack of cardiac reserve.

We propose the use of Flo-Trac/VigileoTM, a semi-invasive technique that estimates cardiac output from the arterial pressure waveform, as a tool for cardiac monitoring during the process of weaning from mechanical ventilation.

References:

1. Richard C and Teboul JL. Weaning failure from cardiovascular origin. Intensive Care Med 2005;31:1605-1607
2. Pinsky MR. Breathing as exercise. Intensive care Med 2000;26:1164-1166
3. Beach T, Millen E, Grenvik A. Hemodynamic response to discontinuation from mechanical ventilation. Crit Care med 1973;1:85-90
4. Lemaire F, Teboul JL, Cinotti L, Giotto G, Abrouk F, Steg G, Macquin-Mavier I and Zapol W. Acute left ventricular dysfunction during unsuccessful weaning from mechanical ventilation. Anesthesiology 1998;69:171-179
5. Jubran A, Mathru M, dries D and Tobin MJ. Continuous recordings from Mixed Venous Oxygen Saturation during Weaning from Mechanical Ventilation and the Ramifications Thereof. Am J Respir Crit Care Med 1998:158:1763-1769
6. De Backer D, El Haddad P, Preiser JC and Vincent JL. Hemodynamic responses to successful weaning from mechanical ventilation after cardiovascular surgery. Intensive Care Med 2000;26:1201-1206
7. Frazier SK et al. Hemodynamic changes during discontinuation of mechanical ventilation in medical intensive care unit patients. Am J Crit Care 2006;15:580-593

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Arterial line in place
* Normal sinus rhythm by electrocardiographic monitoring
* Mechanical ventilation for at least 24 hours
* Ventilation via oral or nasal endotracheal tube
* Patient meets the following weaning criteria before starting weaning protocol:

  * PaO2/FiO2 ratio >200
  * FiO2 equal or less than 50%
  * Positive end-expiratory pressure (PEEP) 5cm H20 or less
  * Respiratory frequency/Tidal volume ratio less 105
  * Respiratory rate < 30 breaths/min
  * Presence of cough and gag reflex
  * 12 hours free from sedation (opioids/benzodiazepine)
  * 2 hours free from sedation in case patient is on Propofol
  * Systolic blood pressure above 90 mmHg and below 180 mmHg
  * Heart rate below 130 beats/min

Exclusion Criteria:

* Known neurological disorder that might impair ventilatory drive
* Known neuromuscular disease
* Inotropic or vasopressor infusion
* Cardiac pacemaker
* Terminal condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients at Memorial Hermann Hospital MICU.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
To describe the hemodynamic changes during the process of discontinuation from mechanical ventilation with the aid of Flo-Trac/Vigileo (TM) | 2 and 9 months

SECONDARY OUTCOMES:
To compare the hemodynamic changes between patients who had successful and those who had unsuccessful discontinuation from mechanical ventilation | 2 and 9 months
To determine if the lack of increase in cardiac output during discontinuation from mechanical ventilation is associated with and predictive of weaning failure | 2 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States